CLINICAL TRIAL: NCT04147234
Title: Phase I, First in Human Trial Evaluating BI 1387446 Alone and in Combination With Ezabenlimab (BI 754091) in Solid Tumors
Brief Title: A Study to Find the Best Dose of BI 1387446 Alone or in Combination With Ezabenlimab (BI 754091) in Patients With Different Types of Advanced or Metastatic Cancer (Solid Tumors)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1426-0001; 2019-001082-32 (EudraCT Number)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Arm A: BI 1387446 50 μg (Experimental): Participants were administered 50 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. The injection volume depended on tumor diameter.
  Interventions: Drug: BI 1387446 50 μg
- Arm A: BI 1387446 100 μg (Experimental): Participants were administered 100 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. The injection volume depended on tumor diameter.
  Interventions: Drug: BI 1387446 100 μg
- Arm A: BI 1387446 200 μg (Experimental): Participants were administered 200 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. The injection volume depended on tumor diameter.
  Interventions: Drug: BI 1387446 200 μg
- Arm A: BI 1387446 400 μg (Experimental): Participants were administered 400 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. The injection volume depended on tumor diameter.
  Interventions: Drug: BI 1387446 400 μg
- Arm B: BI 1387446 50 μg / ezabenlimab 240 mg (Experimental): Participants were administered 50 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. BI 754091 (ezabenlimab) was administered intravenously at the recommended phase II dose of 240 mg once every 3 weeks. The maximum duration of ezabenlimab treatment was 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
  Interventions: Drug: BI 754091
- Arm B: BI 1387446 100 μg / ezabenlimab 240 mg (Experimental): Participants were administered 100 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. BI 754091 (ezabenlimab) was administered intravenously at the recommended phase II dose of 240 mg once every 3 weeks. The maximum duration of ezabenlimab treatment was 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
  Interventions: Drug: BI 754091
- Arm B: BI 1387446 200 μg / ezabenlimab 240 mg (Experimental): Participants were administered 200 μg of BI 1387446 intratumorally under visual inspection for visible skin tumors or under imaging guidance. BI 754091 (ezabenlimab) was administered intravenously at the recommended phase II dose of 240 mg once every 3 weeks. The maximum duration of ezabenlimab treatment was 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
  Interventions: Drug: BI 754091

INTERVENTIONS:
Drug: BI 1387446 50 μg — Participants received 50 μg BI 1387446 intratumorally based on tumor diameter, on Day 1 of a 21-day cycle. Injections were administered under visual inspection for skin tumors or imaging guidance.
  Arms: Arm A: BI 1387446 50 μg
Drug: BI 754091 — Participants received BI 754091 (ezabenlimab) intravenously at a dose of 240 mg once every 21-day cycle.
  Other Names: Ezabenlimab
  Arms: Arm B: BI 1387446 100 μg / ezabenlimab 240 mg; Arm B: BI 1387446 200 μg / ezabenlimab 240 mg; Arm B: BI 1387446 50 μg / ezabenlimab 240 mg
Drug: BI 1387446 100 μg — Participants received 100 μg BI 1387446 intratumorally based on tumor diameter, on Day 1 of a 21-day cycle. Injections were administered under visual inspection for skin tumors or imaging guidance.
  Arms: Arm A: BI 1387446 100 μg
Drug: BI 1387446 200 μg — Participants received 200 μg BI 1387446 intratumorally based on tumor diameter, on Day 1 of a 21-day cycle. Injections were administered under visual inspection for skin tumors or imaging guidance.
  Arms: Arm A: BI 1387446 200 μg
Drug: BI 1387446 400 μg — Participants received 400 μg BI 1387446 intratumorally based on tumor diameter, on Day 1 of a 21-day cycle. Injections were administered under visual inspection for skin tumors or imaging guidance.
  Arms: Arm A: BI 1387446 400 μg

SUMMARY:
This is a study in adults with advanced cancer (solid tumours) in whom previous treatment was not successful. The study tests 2 medicines called BI 1387446 and BI 754091. Both medicines may help the immune system fight cancer. In this study, BI 1387446 is given to humans for the first time.

The purpose of this study is to find out the highest dose of BI 1387446 alone and in combination with BI 754091 the participants can tolerate. BI 1387446 is injected directly into the tumour.

Participants get BI 1387446 injections every week at the beginning and then every 3 weeks.

Some participants get BI 754091 in addition to BI 1387446. BI 754091 is given as an infusion into a vein every 3 weeks.

As long as they benefit from treatment and can tolerate it, participants can stay in the study for up to 2 years and 8 months. During this time, they visit the study site regularly. At these visit, doctors record any unwanted effects. The doctors also regularly check participants' health.

ELIGIBILITY:
Inclusion criteria

* Histologically or cytologically confirmed diagnosis of an advanced, unresectable and/or metastatic malignant solid tumor and indication for treatment
* Patient must have exhausted established treatment options known to prolong survival for the malignant disease, or is not eligible for established treatment options.
* Medically fit and willing to undergo all mandatory trial procedures.
* At least one tumor lesion which is suitable for injection (Screening/initial administration), appropriate for the allocated treatment arm, and measurable.
* At least 1 discrete lesion, in addition to the lesion proposed for injection, which is amenable to biopsy and is not located in the brain, mediastinum or pancreas.
* Adequate organ function or bone marrow reserve
* Further inclusion criteria apply

Exclusion criteria:

* Any investigational or antitumour treatment (including antibodies targeting Programmed Cell Death-1 (PD1) - or programmed Death-Ligand 1 (PDL1)) within 4 weeks or 5 half-life periods (whichever is shorter) prior to the initial administration of BI 1387446 or BI 754091.
* Persistent toxicity from previous treatments (including Immune-related Adverse Events (irAEs)) that has not resolved to ≤ Grade 1, except for alopecia, xerostomia, and immunotherapy related endocrinopathies which may be included if clinically stable on hormone supplements or antidiabetic drugs as per Investigator judgement
* History or evidence of active, non-treatment related autoimmune disease, except for endocrinopathies which may be included if clinically stable on hormone supplements or antidiabetic drugs.
* History or evidence of pneumonitis related to prior immunotherapy
* Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 2 weeks prior to the first dose of BI 1387446 or BI 754091.
* The tumor at the projected injection site has a high risk for local complications, e.g. bleeding related to encasement/infiltration of major blood vessels or contact with liver capsule, compression of vital structures in case of swelling of injected lesion, in the opinion of the Investigator.
* Active infection requiring systemic therapy at the start of treatment in the trial, including active viral hepatitis infection or active tuberculosis infection.
* Cardiac insufficiency New York Heart Association (NYHA) III or IV
* Left ventricular ejection fraction < 50% measured by echocardiography or Multigated Acquisition (MUGA) scan
* Mean resting corrected QT interval (QTc) >470 msec
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona
  - CIO Clara Campal, Madrid
  - Hospital Clínico de Valencia, Valencia
- United Kingdom (3):
  - The Royal Marsden Hospital, Chelsea, London
  - Churchill Hospital, Oxford
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website. The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, multicenter, 2-arm, dose-escalation trial evaluated BI 1387446 administered intratumorally into superficial lesions as a single agent (Arm A) or in combination with intravenous ezabenlimab (Arm B). The primary objectives were to assess safety, determine the maximum tolerated dose for both treatment approaches, and explore preliminary efficacy signals. Patients with progressive disease could cross over to Arm B after completing Cycle 1, provided Arm B is open for recruitment.
Pre-assignment Details: All participants were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the participants) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Arm A: BI 1387446 50 μg: Participants received a 50 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- Arm A: BI 1387446 100 μg: Participants received a 100 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- Arm A: BI 1387446 200 μg: Participants received a 200 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- Arm A: BI 1387446 400 μg: Participants received a 400 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg: Participants received a 50 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
- Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg: Participants received a 100 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
- Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg: Participants received a 200 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
Period: Overall Study
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Started (Started treatment) | 7 | 8 | 7 | 4 | 6 | 3 | 3
Completed (Completed treatment) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 7 | 8 | 6 | 4 | 6 | 3 | 3
Not completed — Clinical deterioration | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Clinical disease progression | 1 | 3 | 1 | 1 | 0 | 1 | 0
Not completed — Objective disease progression | 6 | 4 | 3 | 3 | 5 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication. Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg | Total
Number analyzed (Participants) | 7 | 8 | 7 | 4 | 7 | 5 | 4 | 42
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication. Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover).
  Years
    Arm A: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A | 62.0 (16.6) | 55.3 (10.1) | 65.0 (7.2) | 55.3 (24.4) |  |  |  | 59.7 (14.1)
    Arm B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B |  |  |  |  | 48.6 (14.3) | 57.0 (18.6) | 47.3 (17.5) | 50.9 (16.0)
Sex/Gender, Customized [Number; unit: Participants] — Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover). Population: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication.
  Participants
    Arm A- male: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A- male | 5 | 4 | 3 | 3 |  |  |  | 15
    Arm A- female: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A- female | 2 | 4 | 4 | 1 |  |  |  | 11
    Arm B- male: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B- male |  |  |  |  | 4 | 4 | 2 | 10
    Arm B- female: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B- female |  |  |  |  | 3 | 1 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants] — Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover). Population: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication.
  Participants
    Arm A- Hispanic or Latino: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A- Hispanic or Latino | 0 | 0 | 0 | 0 |  |  |  | 0
    Arm A- Not Hispanic or Latino: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A- Not Hispanic or Latino | 7 | 8 | 7 | 4 |  |  |  | 26
    Arm B- Hispanic or Latino: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B- Hispanic or Latino |  |  |  |  | 1 | 0 | 0 | 1
    Arm B- Not Hispanic or Latino: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B- Not Hispanic or Latino |  |  |  |  | 6 | 5 | 4 | 15
Race/Ethnicity, Customized [Number; unit: Participants] — Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover). Population: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication.
  Participants
    Arm A - Asian: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A - Asian | 0 | 0 | 1 | 0 |  |  |  | 1
    Arm A- Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A- Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 |  |  |  | 1
    Arm A - White: number analyzed (Participants) | 7 | 8 | 7 | 4 | 0 | 0 | 0 | 26
    Arm A - White | 6 | 8 | 6 | 4 |  |  |  | 24
    Arm B - Asian: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B - Asian |  |  |  |  | 0 | 0 | 0 | 0
    Arm B- Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B- Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0 | 0
    Arm B - White: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 16
    Arm B - White |  |  |  |  | 7 | 5 | 4 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response Based on Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1)
Description: Objective response, as defined by the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1), in accordance with Clinical Trial Protocol (CTP) Version 1 and 2, will be presented in terms of the objective response rate (ORR). The ORR is the proportion of patients whose best overall response is a confirmed complete response (CR) or partial response (PR). This determination is based on the investigator's assessment according to RECIST 1.1 criteria, from the date of the first treatment administration until the earliest occurrence of any of the following events: disease progression, death, the last evaluable tumor assessment before the initiation of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
  Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover). Their best overall response is counted, regardless of whether it occurred before or after the crossover.
Time Frame: From start of treatment up to the earliest of progression, death or end of trial (up to 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of any study medication.
  Due to a protocol amendment, only participants who consented under CTP versions 1 and 2 were analyzed for this endpoint. Participants enrolled under CTP version ≥ 3 were assessed using itRECIST and therefore excluded. As a result, the number of participants analyzed for this endpoint is lower than the total in the treated set.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 7 | 8 | 4 | 0 | 7 | 2 | 0
Participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] |  | 0 [0 to 0] | 0 [0 to 0] |

2. Secondary Outcome: Objective Response Based on Response Criteria for Intratumoural Immunotherapy in Solid Tumours (itRECIST)
Description: Objective Response based on Response Criteria for Intratumoural Immunotherapy in Solid Tumours (itRECIST): (CTP version 3 and later) Objective response (OR) by itRECIST will be presented in terms of objective response rate (ORR), which is defined as the rate of patients whose best overall response is confirmed itCR or itPR as determined by the Investigator's assessment according to itRECIST from date of first treatment administration until the earliest of confirmed disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent.
  Cross-over patients are shown in both Arm A (reflecting their initial treatment) and Arm B (reflecting their first treatment post-crossover). Their best overall response is counted, regardless of whether it occurred before or after the crossover.
Time Frame: From start of treatment up to the earliest of progression, death or end of trial (approximately 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of any study medication.
  Due to a protocol amendment, only participants who consented under CTP version ≥ 3 were analyzed for this endpoint. Participants enrolled under CTP versions 1 and 2 were assessed using RECIST 1.1 and therefore excluded. As a result, the number of participants analyzed for this endpoint is lower than the total in the treated set.
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 0 | 0 | 3 | 4 | 0 | 3 | 4
Participants |  |  | 0 [0 to 0] | 1 [0.6 to 80.6] |  | 0 [0 to 0] | 1 [0.6 to 80.6]

3. Secondary Outcome: Best Percentage Change From Baseline in Size of Injected Lesions (CTP Version 1 or 2)
Description: This endpoint evaluated the best percentage change (i.e., greatest reduction) in the size of injected lesions from baseline (the first measurement at the start of treatment) over time. The best percentage change from baseline in the size of injected lesions was analyzed using descriptive statistics.
  All lesion measurements recorded from the start of trial treatment until the earliest of the following were considered: disease progression (assessed under CTP v1 and v2 using RECIST 1.1), initiation of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
  Cross-over patients appear in both Arm A (initial treatment) and Arm B (post-crossover treatment). Their best overall response is counted, regardless of timing.
  Negative values indicate a reduction in injected lesion diameters; positive values indicate an increase.
Time Frame: From start of treatment up to the earliest of progression, death or end of trial (approximately 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of study medication and had both a baseline and at least one post-baseline tumor assessment. Data for this endpoint was collected and evaluated only for participants enrolled under CTP versions 1 and 2 using RECIST 1.1. In these versions, injection of target lesions was not permitted; therefore, injected lesions were collected and assessed separately from target lesions.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 7 | 6 | 2 | 0 | 6 | 2 | 0
Percent change | 23.36 (28.94) | -20.73 (21.95) | -2.78 (3.93) |  | 0.54 (19.24) | 13.33 (18.86) |

4. Secondary Outcome: Best Percentage Change From Baseline in Size of Injected Target Lesions (CTP v3.0 or Later Versions)
Description: This endpoint evaluated the best percentage change (i.e., greatest reduction) in the size of injected target lesions from baseline (the first measurement at the start of treatment) over time. The best percentage change from baseline in the size of injected target lesions was analyzed using descriptive statistics.
  All lesion measurements recorded from the start of trial treatment until the earliest of the following were considered: disease progression (assessed under CTP version 3 and later using itRECIST), initiation of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
  Negative values indicate reduced lesion diameters; positive values indicate increases.
  Cross-over patients are included in Arm A (initial treatment) and Arm B (first post-crossover treatment), with their best response counted regardless of timing.
Time Frame: From start of treatment up to the earliest of progression, death or end of trial (approximately 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of any study medication. Only participants with both a baseline and at least one post-baseline tumor assessment were included in the analysis. Due to a protocol amendment, disease progression for participants consented under CTP version 1 and 2 was assessed using RECIST1.1 and therefore excluded from this endpoint. As a result, the number of participants analyzed is lower than the total number in the treated set.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 0 | 0 | 3 | 4 | 0 | 3 | 4
Percent change |  |  | -6.67 (11.66) | -37.76 (52.67) |  | -17.43 (39.39) | -16.93 (58.42)

5. Secondary Outcome: Best Percentage Change From Baseline in Size of Target Lesions (CTP Version 1 or 2)
Description: This endpoint evaluated the best percentage change (i.e., greatest reduction) in the size of target lesions from baseline (the first measurement at the start of treatment) over time. The best percentage change from baseline in the size of target lesions was analyzed using descriptive statistics.
  All lesion measurements recorded from the start of trial treatment until the earliest of the following were considered: disease progression (assessed under CTP v1 and v2 using RECIST 1.1), initiation of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
  Cross-over patients appear in both Arm A (initial treatment) and Arm B (post-crossover treatment). Their best overall response is counted, regardless of timing.
  Negative values indicate a reduction in lesion diameters; positive values indicate an increase.
Time Frame: From start of treatment until the earliest of progression, death or end of trial (approximately 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of any study medication. Only participants with both a baseline and at least one post-baseline tumor assessment were included in the analysis. Due to a protocol amendment, disease progression for participants consented under CTP version ≥ 3 was assessed using itRECIST and therefore excluded from this endpoint. As a result, the number of participants analyzed is lower than the total number in the treated set.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 7 | 6 | 2 | 0 | 7 | 2 | 0
Percent change | -0.07 (13.92) | 1.02 (6.89) | -0.10 (7.58) |  | 0.07 (13.98) | 0.25 (0.36) |

6. Primary Outcome: Maximum Tolerated Dose (MTD) Based on Number of Dose-limiting Toxicities (DLTs)
Description: The MTD in each arm is defined as the highest dose that is expected to cause less than 25% risk of the true DLT rate being above or equal to 33% during the MTD evaluation period.
  Estimation of the MTD will be based upon the estimation of the posterior probability of the incidence of DLT in toxicity categories during the MTD evaluation period for all evaluable participants.
  The MTD evaluation period is defined as the time from the first administration of any trial medication to the start of the second treatment cycle. Specifically, this is the time from the first dose to either the second administration of ezabenlimab or the fourth administration of BI 1387446, whichever occurs first. If the second dose of ezabenlimab or the fourth dose of BI 1387446 is not given, the evaluation period ends 90 days after the last administration.
Time Frame: From first administration of BI 1387446 until to end of treatment cycle 1 (up to 3 weeks).
Population: The MTD set includes all treated participants evaluable per the clinical trial protocol. This covers those completing required BI 1387446 (and ezabenlimab in Arm B) doses in Cycle 1 and undergoing the Echo/MUGA scan at Cycle 2 Visit 1. Patients stopping due to dose-limiting toxicities are still evaluable. Crossover participants from Arm A to B are included only if evaluable in Arm A. Replaced participants during MTD evaluation are excluded.
Measure: Number; unit: μg (microgram)
Groups:
- Arm A: BI 1387446: Participants received BI 1387446 intratumorally at doses of 50 μg, 100 μg, 200 μg, or 400 μg, depending on tumor diameter. The injections were given under visual inspection for visible skin tumors or under imaging guidance.
- Arm B: BI 1387446 + Ezabenlimab: Participants received BI 1387446 intratumorally at doses of 50 μg, 100 μg, or 200 μg, depending on tumor diameter, along with BI 754091 (ezabenlimab) intravenously at a dose of 240 mg once every 3 weeks. The maximum duration of ezabenlimab treatment was 34 cycles. BI 1387446 injections were preferably administered after completing the ezabenlimab infusion.
Arm/Group | Arm A: BI 1387446 | Arm B: BI 1387446 + Ezabenlimab
Number analyzed (Participants) | 21 | 10
μg (microgram) | NA — The maximum tolerated dose (MTD) was not reached in either treatment arm. According to the Bayesian Logistic Regression Model (BLRM) analysis, all explored dose levels formally met the overdosing criterion, meaning the probability of their dose-limiting toxicity (DLT) rate exceeding 33% was below 25%. | NA — The maximum tolerated dose (MTD) was not reached in either treatment arm. According to the Bayesian Logistic Regression Model (BLRM) analysis, all explored dose levels formally met the overdosing criterion, meaning the probability of their dose-limiting toxicity (DLT) rate exceeding 33% was below 25%.

7. Primary Outcome: Number of Patients With DLT in the MTD Evaluation Period
Description: The MTD evaluation period is defined as the time from the first administration of any trial medication to the start of the second treatment cycle. Specifically, this is the time from the first dose to either the second administration of ezabenlimab or the fourth administration of BI 1387446, whichever occurs first. If the second dose of ezabenlimab or the fourth dose of BI 1387446 is not given, the evaluation period ends 90 days after the last administration.
Time Frame: From first administration of BI 1387446 until to end of treatment cycle 1 (up to 3 weeks).
Population: as for outcome 6
Measure: Number; unit: Number of participants
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 6 | 5 | 6 | 4 | 4 | 3 | 3
Number of participants | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Secondary Outcome: Best Percentage Change From Baseline in Size of Non-injected Target Lesions (CTP v3.0 or Later Versions)
Description: This endpoint evaluated the best percentage change (i.e., greatest reduction) in the size of non-injected target lesions from baseline (the first measurement at the start of treatment) over time. The best percentage change from baseline in the size of non-injected target lesions was analyzed using descriptive statistics.
  All lesion measurements recorded from the start of trial treatment until the earliest of the following were considered: disease progression (assessed under CTP version 3 and later using itRECIST), initiation of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Time Frame: From start of treatment until the earliest of progression, death or end of trial (approximately 1 year).
Population: Treated Set (TS): This set included all participants who received at least one dose of study medication and had both a baseline and at least one post-baseline tumor assessment. Data for this endpoint was collected and evaluated only for participants enrolled under CTP version 3 and later using itRECIST, as these protocol versions allowed injection of target lesions.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm A: BI 1387446 50 μg | Arm A: BI 1387446 100 μg | Arm A: BI 1387446 200 μg | Arm A: BI 1387446 400 μg | Arm B: BI 1387446 50 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 100 μg / Ezabenlimab 240 mg | Arm B: BI 1387446 200 μg / Ezabenlimab 240 mg
Number analyzed (Participants) | 0 | 0 | 3 | 4 | 0 | 3 | 4
Percent change |  |  | -6.23 (6.23) | 1.30 (22.35) |  | 13.42 (14.14) | -17.28 (25.17)

ADVERSE EVENTS:
Time Frame: AE Collection Period: Arm A: From the first BI 1387446 dose until 90 days after the last dose (Residual Effect Period), or until the first Arm B dose, whichever occurred first - for a total duration of up to 14.8 months. Arm B: From the first trial drug dose until 90 days after the last dose (REP), for a total duration of up to 16.4 months. All-Cause Mortality: From the first trial drug dose plus 6 months follow-up after the last dose for a total duration of up to 19.4 months.
Description: Treated set (TS): This patient set includes all patients who were documented to have received at least one dose of any study medication.
  Cross-over patients are depicted both in Arm A (contributing to the patient's initial treatment in Arm A) and Arm B (contributing to the treatment the patient received first after the crossover to Arm B).
Groups:
- BI 1387446 50 ug: Participants received a 50 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- BI 1387446 100 ug: Participants received a 100 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- BI 1387446 200 ug: Participants received a 200 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- BI 1387446 400 ug: Participants received a 400 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. The injection volume was based on tumor diameter.
- BI 1387446 50 ug / Ezabenlimab 240 mg: Participants received a 50 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
- BI 1387446 100 ug / Ezabenlimab 240 mg: Participants received a 100 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
- BI 1387446 200 ug / Ezabenlimab 240 mg: Participants received a 200 μg intratumoral injection of BI 1387446 under visual inspection for visible skin tumors or imaging guidance for non-visible tumors on Day 1 of a 21-day treatment cycle. BI 754091 (ezabenlimab) was administered intravenously at the recommended Phase II dose of 240 mg once every 21-day cycle, with a maximum treatment duration of 34 cycles. BI 1387446 injections were preferably performed after completing the ezabenlimab infusion.
Arm/Group | BI 1387446 50 ug | BI 1387446 100 ug | BI 1387446 200 ug | BI 1387446 400 ug | BI 1387446 50 ug / Ezabenlimab 240 mg | BI 1387446 100 ug / Ezabenlimab 240 mg | BI 1387446 200 ug / Ezabenlimab 240 mg
All-Cause Mortality (participants affected / at risk) | 1/7 | 2/8 | 2/7 | 1/4 | 2/7 | 1/5 | 1/4
Serious Adverse Events (participants affected / at risk) | 2/7 | 4/8 | 3/7 | 0/4 | 5/7 | 2/5 | 2/4
Other Adverse Events (participants affected / at risk) | 6/7 | 8/8 | 7/7 | 4/4 | 7/7 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1387446 50 ug (N=7) | BI 1387446 100 ug (N=8) | BI 1387446 200 ug (N=7) | BI 1387446 400 ug (N=4) | BI 1387446 50 ug / Ezabenlimab 240 mg (N=7) | BI 1387446 100 ug / Ezabenlimab 240 mg (N=5) | BI 1387446 200 ug / Ezabenlimab 240 mg (N=4)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0 | 3 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1387446 50 ug (N=7) | BI 1387446 100 ug (N=8) | BI 1387446 200 ug (N=7) | BI 1387446 400 ug (N=4) | BI 1387446 50 ug / Ezabenlimab 240 mg (N=7) | BI 1387446 100 ug / Ezabenlimab 240 mg (N=5) | BI 1387446 200 ug / Ezabenlimab 240 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1 | 2 | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 3
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 1 | 0 | 2 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal discolouration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Allergic oedema (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 1 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophonesis (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT04147234/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT04147234/SAP_001.pdf